CLINICAL TRIAL: NCT00394849
Title: Effect of Tonsillar Pillar Closure on Postoperative Pain and Bleeding Risk After Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Bruce Matt, Associate Professor, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0006-26
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Hemorrhage; Pain
Keywords: Tonsillectomy; Suturing of tonsillar pillars; pain; postoperative hemorrhage, bleeding
MeSH Terms: conditions — Hemorrhage; Pain; Postoperative Hemorrhage

STUDY DESIGN:
Intervention Model Description: sutured one tonsillar fossa. pain was compared side to side. which side was sutured was randomized
Who Masked: Participant
Masking Description: did not tell participant which side was sutured.
Oversight: Data Monitoring Committee: No

ARMS (2):
- suture one tonsillar fossa (Experimental): Intervention: one tonsillar fossa was sutured. One side was not sutured. Pain was compared side to side.
  Interventions: Procedure: suture one tonsillar fossa
- One side not sutured (No Intervention): Intervention: one tonsillar fossa was sutured. One side was not sutured. Pain was compared side to side.

INTERVENTIONS:
Procedure: suture one tonsillar fossa — one tonsillar fossa was sutured. One side was not sutured. Pain was compared side to side.
  Arms: suture one tonsillar fossa

SUMMARY:
The purpose of this study is to determine if closing the tonsil fossa after tonsillectomy leads to less pain and bleeding risk than leaving it open to heal by secondary intention.

DETAILED DESCRIPTION:
After induction of appropriate general anesthesia, a tonsillectomy was performed and control of bleeding was achieved as is routine for the individual Otolaryngologist performing the procedure. Next the surgeon used 3-0 chromic (absorbable) sutures on tapered needles to close one tonsillar fossa but leave the tonsillar fossa on the other side open. The side chosen was determined by a computer generated schedule. Routine postoperative care was given.

ELIGIBILITY:
Inclusion Criteria:

* Any patient for whom tonsillectomy is recommended for recurrent pharyngitis, obstructive sleep disorder, snoring, halitosis, feeding difficulty associated with adenotonsillar hypertrophy, and who in the investigator's opinion, is capable of providing reliable responses to post-operative follow-up questions as defined in this protocol.

Exclusion Criteria:

* Any patient for whom tonsillectomy is recommended for suspected malignancy or active peritonsillar abscess

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2000-07; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
which side was more painful on or about postoperative day 14 | 14 days
  determined which side was more painful on or about postoperative day 14 by asking patient and/or care giver

SECONDARY OUTCOMES:
Additional information was obtained about details if postoperative bleeding occurred, including which side bled and details of the event | 40 days
  Additional information was obtained about details if postoperative bleeding occurred. Specifically, if postoperative bleeding occurred, we sought to obtain as many details as possible about the events. Items such as when the postoperative bleeding occurred, what was done about it, where the subject was treated, and what the outcome was ( was the bleeding controlled, did the subject have other complications or concerns, etc. were elicited
any other adverse events (complications) | 40 days
  determined if other complications occurred
which side was more painful on or about postoperative day 21 | 21 days
  determined which side was more painful on or about postoperative day 21 by asking patient and/or care giver
overall assessment at the postoperative clinic visit (on or about day 28) | 28 days
  determined overall assessment at the postoperative clinic visit (on or about day 28) by asking patient and/or care giver

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H. Matt, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Childrens' Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matt BH, Krol BJ, Ding Y, Juliar BE. Effect of tonsillar fossa closure on postoperative pain and bleeding risk after tonsillectomy. Int J Pediatr Otorhinolaryngol. 2012 Dec;76(12):1799-805. doi: 10.1016/j.ijporl.2012.09.004. Epub 2012 Sep 25. PMID 23021465